CLINICAL TRIAL: NCT03863301
Title: MRI-guided Single Dose Preoperative Radiotherapy in Low-risk Breast Cancer
Acronym: ABLATIVE-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, HJGD van den Bongard, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL63209 041 18
Record Dates: First submitted 2019-01-15; First posted 2019-03-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm interventional cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided single dose preoperative PBI (Experimental)
  Interventions: Radiation: MR-guided single dose preoperative PBI

INTERVENTIONS:
Radiation: MR-guided single dose preoperative PBI — A single dose of 20Gy to the gross tumor volume (GTV) is prescribed, to the clinical target volume (GTV + 20mm margin) 15Gy is prescribed.

SUMMARY:
This study aims to evaluate the pathologic response at 12 months after single dose preoperative partial breast irradiation in early stage breast cancer patients. Furthermore, the aim is to collect data on response monitoring. Patient-reported outcome measures and treatment-induced toxicity will be evaluated.

DETAILED DESCRIPTION:
In this multi-center single arm interventional cohort study 70 patients will be treated with single dose preoperative partial breast irradiation (PBI). Breast conserving surgery will be performed 12 months following PBI to assess pathologic response. Response monitoring following PBI includes MRI (3T and 7T), liquid biopsies and biopsy of the irradiated tumor.

Results from this trial can change the current treatment of patients with early stage breast cancer. The single dose PBI can be of benefit for all patients who are suitable for postoperative PBI according to current guidelines. If pathologic complete response can be accurately predicted by (one of) the abovementioned response monitoring modalities, the need for surgery will become disputable. Moreover, in patients without expected pathologic complete response, the burden of radiotherapy can be minimized from 3-4.5 weeks of radiotherapy to a single dose of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance scale ≤2.
* Females at least 50 years of age with unifocal cT1N0 breast cancer or females at least 70 years of age with unifocal cT1-2(maximum 3 cm)N0 breast cancer on mammography, ultrasound and MRI.

  * Patients with an indication for chemotherapy or immunotherapy according to Dutch National Oncoline Guidelines or own hospital protocols are not eligible. Patients with an indication for endocrine therapy are eligible.
  * Tumor size as assessed on MRI.
* On tumor biopsy:

  * Bloom-Richardson grade 1 or 2.
  * Non-lobular invasive histological type carcinoma.
  * LCIS or (non-extensive) DCIS is accepted.
  * ER positive tumor receptor.
  * HER2 negative tumor.
* Tumor-negative sentinel node.
* Adequate communication and understanding skills of the Dutch language.

Exclusion Criteria:

* Legal incapacity.
* BRCA1, BRCA2 or CHEK2 gene mutation.
* Previous history of breast cancer or DCIS.
* Other type of malignancy within 5 years before breast cancer diagnosis. Patients with adequately treated malignancy longer than 5 years before breast cancer diagnosis are eligible for inclusion. For adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin no specific time span to breast cancer diagnosis is required for inclusion.
* Collagen synthesis disease.
* Signs of extensive DCIS component on histological biopsy or imaging.
* Invasive lobular carcinoma.
* MRI absolute contraindications as defined by the Department of Radiology.
* Nodal involvement with cytological or histological confirmation.
* Indication for treatment with (neo-)adjuvant chemotherapy.
* Non-feasible dosimetric RT plan.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | up to 12 months
  pCR is assessed 6 or 12 months following single dose radiotherapy. Patients will undergo breast-conserving surgery.

SECONDARY OUTCOMES:
Radiologic response on MRI | up to 12 months
  A 3T MRI will be made 1 week, 3 months, 6 months, 9 months and 12 months following radiotherapy. This will be correlated to the pathologic response.
Biopsy of irradiated tumor | up to 12 months
  A biopsy of the irradiated tumor will be taken before surgery, this will be evaluated for presence of tumor cells. This will be correlated to the pathologic response.
Treatment-induced toxicity | 10 years
  Radiotherapy- and surgery-induced toxicity will be assessed up to 10 years following radiotherapy according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Patient reported outcomes - quality of life | 10 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer-30 (C30), a cancer specific questionnaire on quality of life.
  The C30 consists of the global quality of life (scale 0-100, higher scores indicate higher quality of life), 5 functional domains (physical, role, emotional, cognitive and social functioning, scale 0-100, higher scores indicate better functioning) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties, scale 0-100, higher scores indicate more symptoms). No total score is calculated.
Patient reported outcomes - quality of life | 10 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Breast-23 (BR23), a breast cancer specific questionnaire on quality of life.
  The BR23 consists of 4 functional domains (body image, sexual functioning, sexual enjoyment and future perspectives, scale 0-100, higher scores indicate better functioning) and 4 symptom domains (systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss, scale 0-100, higher scores indicate more symptoms) . No total score is calculated.
Patient reported outcomes - anxiety and depression | 10 years
  Anxiety and depression (Hospital Anxiety and Depression Scale): The scales ranges from 0 to 21 for both domains anxiety and depression separately. Higher scores indicate more complaints of anxiety or depression. No total score is calculated.
Patient reported outcomes - fatigue | 10 years
  Fatigue (Multidimensional Fatigue Index). Five dimensions are present: General fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue. All dimensions range from 4-20, higher scores indicate more symptoms of fatigue on the specific dimension. No total score is calculated.
Patient reported outcomes - work ability | 10 years
  Work ability (Work Ability Index). Seven dimensions are present: current work ability compared to best work ability (scale 0-10), work ability compared to demands of work (scale 2-10), current number of disease (scale 1-7),loss of work ability due to disease (scale 1-6), absenteeism past 12 months (scale 1-5), prognosis work ability in 2 years (scale 1-7), vitality (scale 1-4). A total score of work ability is calculated as the sum of all dimension (scale 7-49). In all dimension higher scores indicate better work ability.
Patient reported outcomes - frailty | 10 years
  Frailty (Groningen Frailty Indicator), one dimension (scale 0-15), higher scores indicate higher level of frailty.
Patient reported outcomes - satisfaction with cosmesis | 10 years
  Satisfaction with cosmesis (questionnaire by Sneeuw et al. and BREAST-Q)). The questionnaire by Sneeuw et al. consists of seven questions, no total score is calculated. These questions are about difference between the treated and untreated breast in terms of size, shape, skin color, firmness and overall cosmesis (scale: no difference, small difference, moderate difference, large difference), visibility of the surgical scar (scale: not distracting, little distracting, quite distracting, very distracting) and satisfaction with the appearance of the treated breast (scale: very satisfied, satisfied, not unsatisfied, unsatisfied, very unsatisfied). No total score is calculated.
  From the BREAST-Q questionnaire only the postoperative domain of satisfaction with the breasts is used (scale 0-100), higher scores indicate more satisfaction.
Local, regional and distant relapse rate | 10 years
  Recurrences up to 10 years following radiotherapy will be evaluated.
Disease free survival | 10 years
  Disease free survival will be evaluated as the interval between treatment and first date of recurrence of disease.
Overall survival | 10 years
  Overall survival will be evaluated as interval between treatment and death.
Tumor infiltrating lymphocytes | up to 12 months
  The presence of tumor infiltrating lymphocytes in the tumor will be assessed at baseline (using the diagnostic biopsy) and following treatment (using the surgical resection). This will be correlated to the pathologic response.
Circulating tumor DNA | up to 12 months
  Patients will be evaluated for the presence of circulating tumor DNA at baseline and following radiotherapy. This will be correlated to the pathologic response.

OTHER OUTCOMES:
Dosimetry of radiotherapy in prone position | 1 month
  Patient can undergo an additional MRI in prone position for a radiotherapy planning study

CONTACTS AND LOCATIONS:
Overall Officials: Desiree van den Bongard, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided